CLINICAL TRIAL: NCT05104918
Title: Vortioxetine as a Novel Anti-depressant With Improvement in Cognitive Abilities - a Randomized Controlled Parallel Assigned Study
Brief Title: Vortioxetine as a Novel Anti-depressant With Improvement in Cognitive Abilities
Acronym: VENUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scotmann Pharmaceuticals (Industry)
Collaborators: Rawalpindi Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VORSCOT
Record Dates: First submitted 2021-10-26; First posted 2021-11-03 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant would be randomly allocated to either of the two interventional groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vorscot Arm (Experimental): Vortioxetine 10 mg
  Interventions: Drug: Vortioxetine
- Vanlafexine Arm (Active Comparator): Venlafaxine 75 mg
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Vortioxetine — 10 mg tablets
  Other Names: VORSCOT tablets
  Arms: Vorscot Arm
Drug: Venlafaxine — 75 mg tablets
  Other Names: Venlafexine
  Arms: Vanlafexine Arm

SUMMARY:
To the best of the knowledge of the Principal Investigators, there was no randomised controlled trial to assess the potential cognitive improvement seen with Vortioxetine, in comparison with some other most commonly used SNRI, when used as directed for the treatment of Major Depressive Disorders. As such the outcome of this trial will provide evidence to assess this claim in the Pakistani population and determine the clinical efficacy when compared to some other commonly used anti-depressants. This would be the first randomized trial dedicated for this assessment in the region with an active control of one of the most commonly used Selective Serotonin and Norepinephrine Reuptake Inhibitors (SSNRIs) in Pakistan for the treatment of depression, Venlafaxine. It can be utilized as an alternative to MDD treatment options, especially where the focus is on improving the cognitive abilities of the patients.

DETAILED DESCRIPTION:
What is Known?

Major Depressive Disorder (MDD) is a distressing and highly prevalent condition which affects the individual's physical, emotional and cognitive well-being, making it one of the leading causes of disability worldwide.

Rationale:

Among the other symptoms, cognitive dysfunctions are one of the major impacts of this disorder and sometimes even overshadow the depressive symptoms2. Disturbances in cognitive functions affect a person's performance in life and work, affecting their concentration, focus, memory, planning, and decision making. Moreover, lack of sleep and dominant-negative thoughts associated with depression also make the cognitive ability worse.

Literature review has consistently demonstrated the negative impact on cognitive abilities affecting the productivity and functioning of individuals with MDD, despite the wide variety of study designs or locations. Cognitive dysfunctions is one of the most common effects reported throughout these studies.

Research gap identified:

Despite the repeated emphasis given in literature indicating the pivotal importance of cognitive abilities on the daily and professional working of humans, this is one domain that is very rarely studied separately in studies.

Relevance, importance, and applicability:

On September 30, 2013, the Food and Drug Administration approved vortioxetine for the treatment of adults with MDD. Vortioxetine's precise mechanism of action is unknown. It is hypothesized that vortioxetine works via blockade of serotonin reuptake; however, vortioxetine is pharmacologically different than other SSRIs because it also works by direct modulation of various serotonin receptors8,9. Chronic therapy with early approved antidepressants causes desensitization of 5-hydroxytryptamine (5-HT1A) on the presynaptic neuron, thereby creating a negative feedback loop and possibly reducing their antidepressive effects. Vortioxetine is an agonist of 5-HT1A on the presynaptic neuron, which can accelerate the antidepressant effects, similar to pindolol, and incorporate serotonin transporter (SERT) blockade10. This molecule acts as an antagonist, agonist, and partial agonist of multiple serotonin receptors and is designed to help reduce depressive symptoms for treatment and maintain response.

Vortioxetine has shown clinically significant results in Major Depressive Disorders (MDD), and possible positive effects on the cognitive abilities of the participants were noted in a few other studies with clinically significant improvement reported. An analysis by Baune et. al showed that Vortioxetine was the only anti-depressant that improved cognitive abilities. Many other studies have backed up this finding of Vortioxetine as an anti-depressant improving the cognitive functions of patients with MDD when taken as directed.

To the best of the knowledge of Principal Investigators, there was no local study done to assess the potential cognitive improvement seen with Vortioxetine when used as directed for the treatment of Major Depressive Disorders.

Purpose of this study:

As such the purpose of this trial is to provide evidence to assess this claim in the Pakistani population. This would be the first randomized trial dedicated for this assessment in the region with active control of one of the most commonly used Selective Serotonin and Norepinephrine Reuptake Inhibitors (SSNRIs) in Pakistan for the treatment of depression, Venlafaxine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Diagnosis of recurrent MDD* > 3 months
3. >26 score of MADRS
4. Participant is a permanent resident of Rawalpindi/Islamabad so that follow up is easy

Exclusion Criteria:

1. Age <18 or >65 years
2. Presence of any other psychiatric disorders (other than MDD)
3. Presence of any organic causes of depression like drug abuse, hypothyroidism, anemia, Cushing syndrome) (Attach reports**)
4. Any physical, cognitive or language disability to perform the cognitive tests
5. Risk of suicide
6. Resistant to previous treatments with either of the interventions (Vortioxetine or Venlafaxine)
7. DSST score >70 at baseline visit

   * According to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) ** Lab tests:

1. Urine drug test for drug abuse 2. Serum TSH to exclude Hypothyroidism 3. Serum Hb to exclude Anaemia 4. Serum Cortisol to exclude Cushing syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 8 weeks
  The MADRS scoring instructions indicate that a total score ranging from 0 to 6 indicates that the patient is in the normal range (no depression), a score ranging from 7 to 19 indicates "mild depression," 20 to 34 indicates "moderate depression," a score of 35 and greater indicates "severe depression," and a total score of 60 or greater indicates "very severe depression."57 There is evidence that an improvement of two points or more on the MADRS is considered clinically relevant.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE Score) | 8 weeks
  The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 25, the result is usually considered to be abnormal (indicating possible cognitive impairment)
Montreal congnitive score | 8 weeks
  Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal. In the initial study data establishing the MoCA, normal controls had an average score of 27.4, compared with 22.1 in people with mild cognitive impairment (MCI) and 16.2 in people with Alzheimer's disease.
Clinical Global Impression (CGI) | 8 weeks
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders.[1] It is a brief 3-item observer-rated scale that can be used in clinical practice as well as in researches to track symptom changes.Its 3 items assess, 1) Severity of Illness (CGI-S), 2) Global Improvement (CGI-I), and 3) Efficacy Index (CGI-E, which is a measure of treatment effect and side effects specific to drugs that were administered.
Digit symbol substitution test (DSST) | 8 weeks
  A score of 400 or higher for the majority of DSST tests is considered passing. The minimum is 200 and the maximum is 600. A score of 400 is comparable to earning a "C" grade on a test which would be considered passing. DSST tests are pass/fail and do not affect student's GPAs.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Umar, Principal Investigator — Rawalpindi Medical College

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- See also: DSST test — https://www.nu.edu/studentservices/testingservices/dantes-subject-standardized-tests-dsst/
- See also: CGI test — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2880930/